CLINICAL TRIAL: NCT07321418
Title: Mid-term Results of Epiphyseal Transfer for Hip Post Septic Epiphyseal Loss. Minimum Five Years Follow-up
Brief Title: Mid-term Results of Epiphyseal Transfer for Hip Post Septic Epiphyseal Loss
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Mostafa Abdelbaky, Resident, Assiut University
Other Study IDs: Mostafa
Record Dates: First submitted 2025-12-12; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Septic Arthritis of the Native Hip; Epiphyseal Arrest, Lower Leg
Keywords: epiphyseal transfer; epiphyseal loss; post septic hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
Absence or loss of the growth plate together with the epiphysis of a long bone presents a very difficult condition to treat. An example of this is the loss of the head and neck of the femur especially as a part of severe sequelae of infantile septic arthritis.

DETAILED DESCRIPTION:
Ever since its advent by Taylor in 1975 , the vascularized fibular free flap has gained popularity and became the gold standard to reconstruct challenging bony defects of the head, neck and extremities. Vascularized fibular flaps offer a great deal of versatility, particularly when reconstructing bony defects larger than 6 cm. In skeletally immature patients, vascularized epiphyseal transfer allows for reconstruction of complex bony defects preserving ongoing longitudinal growth, and provides a reliable articular surface for effective joint function. Although the proximal fibular growth plate is the most popular type of transfer. Therefore, it's mandatory to assess follow up of patients underwent epiphyseal transfer.

Earlier reports of proximal fibular epiphyseal transfer described the use of the peroneal vessels as the pedicle, However the results were overall disappointing and the peroneal artery alone was concluded to be insufficient to support the physeal growth plate. A bipedicled transfer, using the peroneal vessels to support the diaphysis and the anterior tibial vessels or the inferior lateral genicular vessels to support the epiphysis was attempted. Although this showed better outcomes, it was technically more demanding and had a higher risk of complications. Taylor reported the use of the anterior tibial vessels as a single pedicle with success after confirming its role in the blood supply of the fibular diaphysis and epiphysis in a cadaveric study. Another study further popularized the use of the anterior tibial pedicle after introducing the "reverse flow" method and describing the harvest technique. A reported drawback for the use of the anterior tibial pedicle was the occasional need to transect branches of the deep peroneal nerve during the harvest due to their complex relation to the vessels.

This variability in the vascular pedicle employed mandated to the need for a detailed anatomical study of the blood supply of the proximal fibula including the head region, and the supplying vessels, in order to give surgeons appropriate information for choosing the ideal vessel for these complex cases and minimize donor site morbidity. To the best of our knowledge, no such study has been conducted or published in the literature. Moreover, no study has described the anatomic relationship of the deep peroneal nerve branches to the tibialis anterior muscle and their relation to the supplying vessels, which represents another obstacle in the face of popularizing this highly beneficial technique.

Absence or loss of the growth plate together with the epiphysis of a long bone presents a very difficult condition to treat. An example of this is the loss of the head and neck of the femur especially as a part of severe sequelae of infantile septic arthritis. Another example is congenital radial longitudinal deficiency with a previously failed centralization procedure. Management strategies of these and similar problematic conditions are limited and unsatisfactory, with major residual functional disability. Vascularized epiphyseal transfer presents a potential solution to such problems.

ELIGIBILITY:
Inclusion Criteria:

* All cases in Hand and Reconstructive Microsurgery Unit in AUH with epiphyseal transfer for hip post-septic epiphyseal loss.
* Minimum 5 years Follow-up records .

Exclusion Criteria:

* Uncontrolled local infection .
* Patients with incomplete data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: • All cases in Hand and Reconstructive Microsurgery Unit in AUH with epiphyseal transfer for hip post-septic epiphyseal loss.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional outcome of the hip. | 5 years
  • Bone union will be evaluated according to de Boer et al in 1989
functional outcome | 5 years
  The Oxford Hip Score (OHS) for hip function